CLINICAL TRIAL: NCT05350033
Title: Transcranial Direct Current Stimulation on Inhibitory Control in Addictions: a Triple-blinded, Sham-controlled Clinical Trial.
Brief Title: Transcranial Direct Current Stimulation on Inhibitory Control in Addictions.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad de Almeria (Other)
Collaborators: Junta de Andalucia (Other Government)
Responsible Party: Principal Investigator, Fernando Sanchez-Santed, Professor, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TESADIC
Record Dates: First submitted 2022-03-14; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Substance-Related Disorders
Keywords: substance abuse; transcraneal electrical stimulation; tDCS; inhibitory control; drug craving; treatment adherence
MeSH Terms: conditions — Substance-Related Disorders; Treatment Adherence and Compliance | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: * Group 1: Active-stimulation in Phase 1 and Phase 2
  * Group 2: Active-stimulation in Phase 1 and Sham-stimulation in Phase 2
  * Group 3: Sham-stimulation in Phase 1 and Active-stimulation in Phase 2
  * Group 4: Sham-stimulation in Phase 1 and Phase 2
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Care providers communicate to the PI for participants' availability each week. PI assigns an anonymization code that serves to activate the stimulation device in active or sham-mode, blinded to investigators or participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active-Active (Experimental): Participants will receive active-tDCS stimulation (anode F4 / cathode F3) at 2 mA during 20 min in Phase 1 (5 sessions, intersession time-24h) and in Phase 2 (5 sessions, intersession time-24h).
  Interventions: Device: tDCS - tDCS
- Active-Sham (Experimental): Participants will receive active-tDCS stimulation (anode F4 / cathode F3) at 2 mA during 20 min in Phase 1 (5 sessions, intersession time-24h), and sham-tDCS at 2 mA (active-stimulation lasting for 1 min) in Phase 2 (5 sessions, intersession time-24h).
  Interventions: Device: tDCS - Sham
- Sham-Active (Experimental): Participants will receive sham-tDCS stimulation (anode F4 / cathode F3) at 2 mA (active-stimulation lasting for 1 min) in Phase 1 (5 sessions, intersession time-24h), and active-tDCS at 2 mA during 20 min in Phase 2 (5 sessions, intersession time-24h).
  Interventions: Device: Sham - tDCS
- Sham-Sham (Sham Comparator): Participants will receive sham-tDCS stimulation (anode F4 / cathode F3) at 2 mA (active-stimulation lasting for 1 min) in Phase 1 (5 sessions, intersession time-24h), and sham-tDCS at 2 mA (active-stimulation lasting for 1 min) in Phase 2 (5 sessions, intersession time-24h).
  Interventions: Device: Sham - Sham

INTERVENTIONS:
Device: tDCS - tDCS — active-tDCS administered during 10 sessions, in Phase 1 and Phase 2
  Arms: Active-Active
Device: tDCS - Sham — active-tDCS administered during 5 sessions, in Phase 1
  Arms: Active-Sham
Device: Sham - tDCS — active-tDCS administered during 5 sessions, in Phase 2
  Arms: Sham-Active
Device: Sham - Sham — sham-tDCS administered during 10 sessions, in Phase 1 and Phase 2
  Arms: Sham-Sham

SUMMARY:
The research in neuroscience of the last 20 years is defined, in addition to continuing to advance in the field of behavioral and pharmacological therapy, by the birth and development of a new therapeutic category, called neuromodulation. Neuromodulation offers the possibility of producing changes in the Nervous System (SN) and therefore, in behavior, in addition to lasting over time. One of the most used non-invasive neuromodulation techniques is transcranial direct current stimulation (tDCS). The benefits of tDCS are promising and varied, so it is a potential neurorehabilitation tool, which has also shown its greatest effectiveness when accompanied by complementary rehabilitation treatment. The present study focuses on the effect of tDCS on addiction. Specifically, there is a great problem with the high rates of relapse presented by those individuals who try to abandon addictive behavior. Therefore, the maintenance of the abstinence period is the central theme of addiction research and the main challenge of rehabilitation at present. For that aim, the intervention will be carried out in a sample in the intermediate phase (internal) in the NOESSO (No EstáS Sólo) therapeutic community (Almería, Spain), between day 15 after arrival and the first day to leave on leave (day 45-60). The research will be made up of a previous period of selection and collection of data related to addiction, together with two phases or moments of correlative intervention and evaluation. Users will receive a bilateral (F3/F4) and repeated stimulation of 2 mA intensity for 20 min each, that is, every 24h for 5 consecutive days in each phase. Through this procedure, the aim is to seek to increase adherence to treatment in the early intervention phase and decrease the dropout rate due to the enhancement of inhibitory control. On the other hand, in the second phase, advanced intervention is sought to reduce craving, through an improvement in inhibitory and emotional control at the time of returning to the context of real consumption. In order to increase the knowledge about intra-individual differences in the effect of tDCS, researchers will compare the early intervention (Phase 1, at the begging of the rehabilitation process) with the advanced intervention (Phase 2, right before the first leave).

DETAILED DESCRIPTION:
The research in behavioral neuroscience of the last 20 years is defined, in addition to continuing to advance in the field of behavioral and pharmacological therapy, by the birth and development of a new therapeutic category, called neuromodulation. Neuromodulation, especially non-invasive neuromodulation, has had a great impact on the current scientific landscape, encompassing the participation and interest of different disciplines such as medicine, bioengineering, psychology, and neuroscience. Scientific publications, as well as the media impact of this type of technique, have been increasing and continue to grow today. Neuromodulation offers the possibility of producing changes in the Nervous System (SN), and these also last over time. These techniques were born with the idea of avoiding the side effects of pharmacological therapy while offering a direct impact on the improvement of pathological symptoms. The changes produced by neuromodulation are promoted, among others, by ultrasound, microscale magnetic fields, and electricity. This last resource, electrical energy, is used by electrical neuromodulation techniques, one of the most studied branches of neuromodulation currently. Electrical neuromodulation starts from the basis that the neurons of our SN communicate with each other through chemical and electrical processes. By applying low-intensity electricity directly to the SN, it is possible to modulate the neuronal communication of the stimulated area by increasing or decreasing the excitability of the membrane of the target neuron field. Electrical neurostimulation encompasses different techniques, among which is Transcranial Direct Current Stimulation (tDCS). The present project focuses on tDCS since it is the technique that has demonstrated higher success rates as well as fewer, or no, side effects.

The tDCS consists of a device that contains a ≈9-volt battery. Two electrodes generally emanate from this device: the anode (positive pole), and the cathode (negative pole). Once placed non-invasively on the scalp, electricity flows between both electrodes at very low intensity (maximum 2 mA) for an approximate time of 20 minutes. This flow is barely noticeable to the user, who usually feels only a slight itch in the area of the electrodes that disappear after 60 seconds. However, under the skull, in the brain, electrical changes occur in the neurons in the area. Usually, under the anode there is a depolarization of the neuronal membrane, generating excitability, that is, the first step to greater activity. Under the cathode, most of the time, the opposite process occurs, a polarization that precedes a neuronal inhibition. This change in activity has been recorded by different studies and methods, directly measuring the change in cortical excitability, oxyhemoglobin level, white matter or the change in the levels of neurotransmitters such as gamma-aminobutyric acid (GABA) and Glutamate.

So far, tDCS has proven to be an effective yet safe technique, including relatively simple use causing the least discomfort to the user. The most common side effect that has been recorded is the slight itching in the area of the electrodes that also decreases after 60 seconds. This sensation can be controlled and reduced by using an adequate amount of conductive fluid, as well as by greater separation between both electrodes. In fact, tDCS has been shown to be a safe technique for use in children, adolescents, and older people. Administration of tDCS has been shown not to change indirect biomarkers of brain damage (N-acetyl-asperate), as well as levels of other related metabolites. In addition, no adverse effects on cardiac function have been found from stimulation and no convulsive effects have been associated with tDCS. However, to ensure effective and safe stimulation, possible skin sensitivity, medication, substance use, psychiatric disorders or a history of epilepsy should be recorded for each participant, thus controlling their possible interaction. A recent study conducted an updated tDCS safety exploration with more than 1,000 subjects, including participants from vulnerable populations, with an application of more than 33,200 sessions of tDCS, with stimulation of up to 4 mA and up to 40 minutes per session. The results showed no evidence of any serious adverse effects or irreversible damage.

The interesting thing about tDCS is not only the direct changes it produces on brain activity but those it produces directly on behavior and are perceptible. In a recent review on tDCS conducted by our research team, it was found that tDCS produces beneficial effects on human motor function when the motor cortex and cerebellum are stimulated. In addition, it has been found that the application of tDCS can reduce neuropathic pain, improve psychopathologies such as depression, schizophrenia and anxiety, as well as improving cognitive processes such as learning, perception and memory. The benefits of tDCS are promising and varied, so it is a potential neurorehabilitation tool, which has also shown its greatest effectiveness when accompanied by complementary rehabilitation treatment.

The excitatory or inhibitory effect of a single session of tDCS has been shown to last up to 90 minutes after stimulation. However, what makes this neurorehabilitation technique really interesting is its long-term effect. It has been proven that when stimulation is performed continuously, in repeated sessions, there is a therapeutic benefit that has been maintained up to 3 months after the last stimulation session. In fact, the alteration produced by tDCS in the glutamatergic system has been shown to be related to an increase in brain-derived neurotrophic factor (BDNF), a key molecule for synaptic plasticity. That is, there are changes in the brain that last over time.

tDCS and addiction The present study focuses on the effect of tDCS on addiction. Substance addiction is one of the most important mental health problems today. Specifically, there is a great problem with the high rates of relapse presented by those individuals who try to abandon addictive behavior. Therefore, the maintenance of the abstinence period is the central theme of addiction research and the main challenge of rehabilitation in the present. In this line, it has been found that stimulating through tDCS areas related to the circuits of addiction and decision making, preferably the dorsolateral prefrontal cortex (DLPFC) has been possible to modulate the processes of addiction. Anodal stimulation with tDCS over DLPFC has been shown to improve cognitive processes, such as working memory and decision making. This is because this brain area is involved in key processes of addiction, such as impulse control and stimulus salience. Neuroimaging studies have shown that DLPFC dysfunction is related, in addition to these processes, directly to compulsive drug use. To date, stimulation of this brain region has been found to decrease craving for the substance of addiction, relapse rate, and level of substance use such as alcohol, tobacco, cocaine and methamphetamine. Therefore, tDCS is presented as a potential rehabilitation tool that can produce great benefits for addiction, especially in the withdrawal phase, preventing relapse.

In addition to addiction-related behaviors, such as craving, relapse, and the emotions that accompany addiction, such as depressive or anxiety symptoms, the present study aims to deeply analyze the psychological process underlying addiction: inhibitory control. Inhibitory control is the ability to contain or stop an inappropriate behavior or response, and its alteration leads to maladaptive behaviors such as impulsivity and compulsivity. Previous studies have found a direct relationship between addiction and high impulsivity, high compulsivity, and a preference for risky decision-making. With tDCS, it has been possible to improve impulsivity and compulsivity, not only in addiction, but also in behaviors related, such as pathological gambling and binge eating disorders.

Although there are increasingly consolidated literature on the therapeutic benefits of tDCS applied to DLPFC (F3/F4) on addiction, the latest review on tDCS and addiction points out the need to study its effect on polyaddiction to different substances, which constitutes a population much closer to reality, addiction to a single substance being uncommon. In addition, it is postulated that the samples used in tDCS studies are too small. Finally, a determining limitation is that the opportune moment to apply tDCS is not yet known, if in a more initial phase of addiction rehabilitation, or in a later phase when the rehabilitation process is in a more advanced state. Therefore, this study aims to cover in a longitudinal study an important sample of people with polyaddiction treated in their therapeutic context, to verify the effects of tDCS on the direct components of addiction, such as craving and relapse, as well as on the basic psychological process that underlies addiction: inhibitory control. The intervention will be applied in the initial phase of rehabilitation, as well as in an advanced phase of it. Through the sham condition of tDCS, a control group will be created. All patients will participate in an intervention program while receiving tDCS treatment. This procedure aims to study the efficacy of tDCS for the improvement of inhibitory control and addiction in a process of addiction rehabilitation.

It is expected, therefore, that through the neuromodulation of inhibitory control through the application of tDCS in DLPFC there will be a benefit in the rehabilitation of a population with polyaddiction, which is reflected in greater control of the levels of impulsivity and compulsiveness, better decision making, and therefore, lower rates of anxiety, craving for the substance, relapse rate and an increase in quality of life.

This project is proposed in collaboration and close coordination with the NOESSO (No EstáS Sólo) Association. NOESSO is dedicated, as a non-profit association, to the reception and treatment of people with addictions. It is integrated into the healthcare network for the treatment of addiction of the Junta de Andalucía, in Spain. It is composed of various rehabilitation and integration centers in the province of Almeria. In Laujar de Andarax there is located the center of primary rehabilitation reception (Cortijo La Quita Therapeutic Community), where patients referred from various centers are admitted. The rehabilitation process follows a strict protocol, in accordance with national and regional guidelines, which combines a multidisciplinary strategy. After the first period of detoxification of a minimum of 15 days, the patient enters a therapeutic program where doctors, psychologists, educators, and social workers work according to an individualized program. The rehabilitation process is completed with a progressive program of departures from the center so that patients gradually face their previous environment. The first departure occurs between 45 and 60 days after admission, at the discretion of the clinical team. NOESSO receives between 90-100 admissions annually. Of these, between 15-20% reach therapeutic discharge, and 25-30% achieve partially achieve objectives. They voluntarily abandon between 20-25% and the rest enter other casuistries without therapeutic success. Therefore, the percentage of dropouts and relapses is high. In fact, in the first scheduled departure from the center, about 20% of relapses are recorded, objectified by control of substances by urinalysis.

Hypothesis: Through the neuromodulation of inhibitory control through the application of tDCS in DLPFC there will be a benefit in the rehabilitation of a population with polyaddiction, which is reflected in greater control of the levels of impulsivity and compulsiveness, better decision making, and therefore, lower rates of anxiety, craving for the substance, relapse rate and an increase in quality of life.

General objective: to reduce the relapse rate, thus increasing the success rate, and increasing the quality of life of patients undergoing a rehabilitation process for substance addiction.

The objectives of this project are aimed at improving the inhibitory control of patients with polyaddiction through the repeated application of stimulation with tDCS. It is expected that the consequence of this improvement will be reflected in greater adherence to treatment, that is, in a significant reduction in the rate of relapse and abandonment. The objectives, therefore, can be divided into three different categories, although all of them are interrelated. Throughout the four evaluations that will be carried out (pre and post of each phase), the objective is to induce a progressive improvement of all the components of inhibitory control that will be measured by neurobehavioral tasks. That is, the goal is for participants who receive tDCS to show a lower rate of risky decisions, i.e. a higher Net Score in the Iowa Gambling Task and a lower number of false alarms in the Go/No Go task. It is expected for participants who have received tDCS to show lower scores on the compulsivity (MOCI) and impulsivity (BIS-11) questionnaires, as well as a better emotional state reflected in more favorable scores on symptoms of depression (BDI-BECK), anxiety (STAI-E/R), fatigue (VAS) and consequently, a higher score on the perceived quality of life (WHOQOL-BREF). The change that treatment with tDCS can suppose on these variables is expected to be reflected in the primary objective of this work, which is the reduction of substance craving (VAS), and therefore, greater adherence to treatment, reflected in a lower relapse rate and a greater number of patients who do not abandon therapy. These changes produced in a population with polyaddiction will be a novelty in the panorama of the scientific literature regarding neuromodulation, since to date there is still a demand for studies on tDCS in the rehabilitation of several substances, a situation closer to the reality of this health problem.

ELIGIBILITY:
Inclusion Criteria:

* Substance abuse
* Under clinical treatment at the Noesso Addiction Rehabilitation Center La Quinta, Laujar de Andarax, Spain
* Participation approved by the clinical team
* Participation approved by the experimental team by means of the Göttingen screening questionnaire
* Signed informed consent
* At least 26 points in the Montreal Cognitive Assessment (MOCA) evaluation

Exclusion Criteria:

* Epilepsy or history of epilepsy (convulsions due compsumtion not included)
* Cardiopathy or cardiac electronic devices
* Skin reaction or high sensitivity to tDCS
* Head metallic implant
* Serious mental disease
* Exclusion because of clinical criteria (physician, psychologist)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Dropouts phase 1: participants that abandon the treatment phase | 45-60 days
  Number of participants that abandon the treatment phase before the first free weekend outside the center
Dropouts phase 2: participants that abandon the treatment after the first free weekend outside the center | 47-62 days
  Number of participants that abandon the treatment after the first free weekend outside the center
Relapses: | 41-62 days
  Number of relapses on drug comsuption during the first free weekend outside the center

SECONDARY OUTCOMES:
VAS - Craving | Daily during the total ten days of intervention
  Quantification fo drug craving by Visual Analogue Scale (VAS): This is a visual analog scale, which means that it does not present lexical items. On the contrary, the user only has to mark on the scale from 0 to 10 the degree of a perceived sensation or state of health, in this case the desire for drug (craving)
VAS - Fatigue | For each interventional phase: first and fifth day
  Quantification fo drug craving by Visual Analogue Scale (VAS): This is a visual analog scale, which means that it does not present lexical items. On the contrary, the user only has to mark on the scale from 0 to 10 the degree of a perceived sensation or state of health, in this case fatigue.
STAI-E/R | For each interventional phase: first and fifth day
  Questionnaire of anxiety state / trait STAI-E / R, is one of the most used tests to measure anxiety, since it allows to differentiate between the stable anxiety in the own time of people with threatening attribution to a wide range of situations, and the anxiety that occurs at that specific moment or transitory emotional state, that the subject is conscious.
WHOQOL-BREF | For each interventional phase: first and fifth day
  WHOQOL-BREF is the Spanish version of the most used test in the field of health to evaluate quality of life in a generic and self-reported way. It consists of 26 items, classified into 4 dimensions (physical, psychological, social relations and environment). It is fast and effective, however it does not allow specific clinical areas to be evaluated in a concrete way.
Beck BDI-BECK | For each interventional phase: first and fifth day
  Beck BDI-BECK-II inventory is widely used to assess the degree of depression. It consists of 21 items indicative of symptoms such as sadness, crying, loss of pleasure, guilt, and desire for suicide according to the Diagnostic and Statistical Manual of Mental Disorders (DSM). Its administration is self-report and provides a measure of presence and severity in adults and adolescents. It is indicated for clinical psychology, neuropsychology, and forensics.
BIS-11 | For each interventional phase: first and fifth day
  Barratt impulsivity scale (BIS-11). It evaluates impulsivity and its subtypes: cognitive impulsivity, motor impulsivity and impulsivity related to non-planning. The scale consists of 30 Likert-type items and its administration is self-reported. This scale is widely applied in research related to clinical population and substance abuse.
MOCI | For each interventional phase: first and fifth day
  Maudsley Obsessional-Compulsive Inventory (MOCI) (Spanish version). It evaluates compulsivity and its subtypes: (a) checking, (b) cleanliness, (c) slowness and repetition, and (d) doubt and awareness. It has been developed in order to investigate the traits of compulsivity. The questionnaire comprises 30 items with true/false answers. The results are interpreted as a measure of the intensity of compulsive behaviors since the high false alarms in the Go/no-go task are related to a high score in the MOCI questionnaire.
IGT | For each interventional phase: first and fifth day
  Iowa Gambling Task (IGT): is a neurobehavioral task that measures risky decision-making. Four decks of cards will appear on the computer screen. Each participant will have to choose a card from any deck by clicking on it. The task will consist of 100 essays. In each choice, decks A and B will generate a profit of 100 points and decks C and D of 50 points. However, every 10 trials the choice of the first deck will result in a net loss of 250 points, while the choice of the second will result in a net gain of the same amount. All participants will start with 2000 points and will be instructed to maximize their profits.
  The main variable Net Score: is the total score obtained by the participant. People with a low Net Score have shown a deficit in performing this task, such as people with substance addiction.
Go/no-go | For each interventional phase: first and fifth day
  Go/no-go task has been widely used to assess cognitive control, compulsion, and inhibitory control of behavior. A recently published version by our research group will be used. It consist of the presentation of circles of two different colors separated by a fixing point, during 200 tests. What participants should do is respond by pressing the computer's keyboard space bar as quickly as possible if the circle that appears is green (Go test), and avoid responding to the appearance of blue circles (No-Go test). 80% of the trials will be Go trials. Both stimuli will appear on the screen for 350ms. The presentation time will be adjusted to the participant's reaction time (+50ms or -50ms). The interval between stimuli will be variable, between 800ms and 1500ms. The main variable is "false alarms", pressing the key in No-Go trials.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Sánchez-Santed, PhD, Principal Investigator — Universidad de Almeria
Locations (1):
- Psychobiology Lab, Almería, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected Individual Participants Data (IPD) will be shared in .csv files together with readme.txt files describing data processing
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available between six and twelve months after each potential publication
Access Criteria: No restrictions will be applied

REFERENCES:
- [Background] Salling MC, Martinez D. Brain Stimulation in Addiction. Neuropsychopharmacology. 2016 Nov;41(12):2798-2809. doi: 10.1038/npp.2016.80. Epub 2016 May 31. PMID 27240657
- [Background] Bajbouj M, Padberg F. A perfect match: noninvasive brain stimulation and psychotherapy. Eur Arch Psychiatry Clin Neurosci. 2014 Nov;264 Suppl 1:S27-33. doi: 10.1007/s00406-014-0540-6. Epub 2014 Sep 25. PMID 25253645
- [Background] Page SJ, Cunningham DA, Plow E, Blazak B. It takes two: noninvasive brain stimulation combined with neurorehabilitation. Arch Phys Med Rehabil. 2015 Apr;96(4 Suppl):S89-93. doi: 10.1016/j.apmr.2014.09.019. PMID 25813373
- [Background] Hsu TY, Juan CH, Tseng P. Individual Differences and State-Dependent Responses in Transcranial Direct Current Stimulation. Front Hum Neurosci. 2016 Dec 21;10:643. doi: 10.3389/fnhum.2016.00643. eCollection 2016. PMID 28066214
- [Background] Dubljevic V, Saigle V, Racine E. The rising tide of tDCS in the media and academic literature. Neuron. 2014 May 21;82(4):731-6. doi: 10.1016/j.neuron.2014.05.003. PMID 24853934
- [Background] Lewis PM, Thomson RH, Rosenfeld JV, Fitzgerald PB. Brain Neuromodulation Techniques: A Review. Neuroscientist. 2016 Aug;22(4):406-21. doi: 10.1177/1073858416646707. Epub 2016 Apr 29. PMID 27130839
- [Background] De Ridder D, Perera S, Vanneste S. State of the Art: Novel Applications for Cortical Stimulation. Neuromodulation. 2017 Apr;20(3):206-214. doi: 10.1111/ner.12593. Epub 2017 Mar 28. PMID 28371170
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] McKendrick R, Parasuraman R, Ayaz H. Wearable functional near infrared spectroscopy (fNIRS) and transcranial direct current stimulation (tDCS): expanding vistas for neurocognitive augmentation. Front Syst Neurosci. 2015 Mar 9;9:27. doi: 10.3389/fnsys.2015.00027. eCollection 2015. PMID 25805976
- [Background] Zheng X, Schlaug G. Structural white matter changes in descending motor tracts correlate with improvements in motor impairment after undergoing a treatment course of tDCS and physical therapy. Front Hum Neurosci. 2015 Apr 30;9:229. doi: 10.3389/fnhum.2015.00229. eCollection 2015. PMID 25983684
- [Background] Kim S, Stephenson MC, Morris PG, Jackson SR. tDCS-induced alterations in GABA concentration within primary motor cortex predict motor learning and motor memory: a 7 T magnetic resonance spectroscopy study. Neuroimage. 2014 Oct 1;99:237-43. doi: 10.1016/j.neuroimage.2014.05.070. Epub 2014 Jun 3. PMID 24904994
- [Background] Bachtiar V, Near J, Johansen-Berg H, Stagg CJ. Modulation of GABA and resting state functional connectivity by transcranial direct current stimulation. Elife. 2015 Sep 18;4:e08789. doi: 10.7554/eLife.08789. PMID 26381352
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Background] Minhas P, Datta A, Bikson M. Cutaneous perception during tDCS: role of electrode shape and sponge salinity. Clin Neurophysiol. 2011 Apr;122(4):637-8. doi: 10.1016/j.clinph.2010.09.023. Epub 2010 Nov 12. No abstract available. PMID 21075048
- [Background] Moliadze V, Antal A, Paulus W. Electrode-distance dependent after-effects of transcranial direct and random noise stimulation with extracephalic reference electrodes. Clin Neurophysiol. 2010 Dec;121(12):2165-71. doi: 10.1016/j.clinph.2010.04.033. Epub 2010 Jun 15. PMID 20554472
- [Background] Aree-uea B, Auvichayapat N, Janyacharoen T, Siritaratiwat W, Amatachaya A, Prasertnoo J, Tunkamnerdthai O, Thinkhamrop B, Jensen MP, Auvichayapat P. Reduction of spasticity in cerebral palsy by anodal transcranial direct current stimulation. J Med Assoc Thai. 2014 Sep;97(9):954-62. PMID 25536713
- [Background] Cosmo C, Baptista AF, de Araujo AN, do Rosario RS, Miranda JG, Montoya P, de Sena EP. A Randomized, Double-Blind, Sham-Controlled Trial of Transcranial Direct Current Stimulation in Attention-Deficit/Hyperactivity Disorder. PLoS One. 2015 Aug 12;10(8):e0135371. doi: 10.1371/journal.pone.0135371. eCollection 2015. PMID 26267861
- [Background] Krishnan C, Santos L, Peterson MD, Ehinger M. Safety of noninvasive brain stimulation in children and adolescents. Brain Stimul. 2015 Jan-Feb;8(1):76-87. doi: 10.1016/j.brs.2014.10.012. Epub 2014 Oct 28. PMID 25499471
- [Background] Floel A, Suttorp W, Kohl O, Kurten J, Lohmann H, Breitenstein C, Knecht S. Non-invasive brain stimulation improves object-location learning in the elderly. Neurobiol Aging. 2012 Aug;33(8):1682-9. doi: 10.1016/j.neurobiolaging.2011.05.007. Epub 2011 Jun 17. PMID 21684040
- [Background] Rango M, Cogiamanian F, Marceglia S, Barberis B, Arighi A, Biondetti P, Priori A. Myoinositol content in the human brain is modified by transcranial direct current stimulation in a matter of minutes: a 1H-MRS study. Magn Reson Med. 2008 Oct;60(4):782-9. doi: 10.1002/mrm.21709. PMID 18816828
- [Background] Vandermeeren Y, Jamart J, Ossemann M. Effect of tDCS with an extracephalic reference electrode on cardio-respiratory and autonomic functions. BMC Neurosci. 2010 Mar 16;11:38. doi: 10.1186/1471-2202-11-38. PMID 20233439
- [Background] Tanaka S, Watanabe K. [Transcranial direct current stimulation--a new tool for human cognitive neuroscience]. Brain Nerve. 2009 Jan;61(1):53-64. Japanese. PMID 19177807
- [Background] Bikson M, Datta A, Elwassif M. Establishing safety limits for transcranial direct current stimulation. Clin Neurophysiol. 2009 Jun;120(6):1033-4. doi: 10.1016/j.clinph.2009.03.018. Epub 2009 Apr 24. No abstract available. PMID 19394269
- [Background] Bikson M, Grossman P, Thomas C, Zannou AL, Jiang J, Adnan T, Mourdoukoutas AP, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Jankord R, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Safety of Transcranial Direct Current Stimulation: Evidence Based Update 2016. Brain Stimul. 2016 Sep-Oct;9(5):641-661. doi: 10.1016/j.brs.2016.06.004. Epub 2016 Jun 15. PMID 27372845
- [Background] Sanchez-Kuhn A, Perez-Fernandez C, Canovas R, Flores P, Sanchez-Santed F. Transcranial direct current stimulation as a motor neurorehabilitation tool: an empirical review. Biomed Eng Online. 2017 Aug 18;16(Suppl 1):76. doi: 10.1186/s12938-017-0361-8. PMID 28830433
- [Background] Mehta S, McIntyre A, Guy S, Teasell RW, Loh E. Effectiveness of transcranial direct current stimulation for the management of neuropathic pain after spinal cord injury: a meta-analysis. Spinal Cord. 2015 Nov;53(11):780-5. doi: 10.1038/sc.2015.118. Epub 2015 Jul 21. PMID 26193817
- [Background] Nitsche MA, Boggio PS, Fregni F, Pascual-Leone A. Treatment of depression with transcranial direct current stimulation (tDCS): a review. Exp Neurol. 2009 Sep;219(1):14-9. doi: 10.1016/j.expneurol.2009.03.038. Epub 2009 Apr 5. PMID 19348793
- [Background] Brunelin J, Mondino M, Gassab L, Haesebaert F, Gaha L, Suaud-Chagny MF, Saoud M, Mechri A, Poulet E. Examining transcranial direct-current stimulation (tDCS) as a treatment for hallucinations in schizophrenia. Am J Psychiatry. 2012 Jul;169(7):719-24. doi: 10.1176/appi.ajp.2012.11071091. PMID 22581236
- [Background] Batista EK, Klauss J, Fregni F, Nitsche MA, Nakamura-Palacios EM. A Randomized Placebo-Controlled Trial of Targeted Prefrontal Cortex Modulation with Bilateral tDCS in Patients with Crack-Cocaine Dependence. Int J Neuropsychopharmacol. 2015 Jun 10;18(12):pyv066. doi: 10.1093/ijnp/pyv066. PMID 26065432
- [Background] Sanchez-Kuhn A, Perez-Fernandez C, Moreno M, Flores P, Sanchez-Santed F. Differential Effects of Transcranial Direct Current Stimulation (tDCS) Depending on Previous Musical Training. Front Psychol. 2018 Sep 10;9:1465. doi: 10.3389/fpsyg.2018.01465. eCollection 2018. PMID 30250439
- [Background] Costa TL, Lapenta OM, Boggio PS, Ventura DF. Transcranial direct current stimulation as a tool in the study of sensory-perceptual processing. Atten Percept Psychophys. 2015 Aug;77(6):1813-40. doi: 10.3758/s13414-015-0932-3. PMID 26139152
- [Background] Javadi AH, Cheng P. Transcranial direct current stimulation (tDCS) enhances reconsolidation of long-term memory. Brain Stimul. 2013 Jul;6(4):668-74. doi: 10.1016/j.brs.2012.10.007. Epub 2012 Oct 31. PMID 23137702
- [Background] Zhao S, Dou Z, Wei X, Li J, Dai M, Wang Y, Yang Q, He H. Task-concurrent anodal tDCS modulates bilateral plasticity in the human suprahyoid motor cortex. Front Hum Neurosci. 2015 Jun 24;9:370. doi: 10.3389/fnhum.2015.00370. eCollection 2015. PMID 26157383
- [Background] Grecco LA, Duarte Nde A, de Mendonca ME, Pasini H, Lima VL, Franco RC, de Oliveira LV, de Carvalho Pde T, Correa JC, Collange NZ, Sampaio LM, Galli M, Fregni F, Oliveira CS. Effect of transcranial direct current stimulation combined with gait and mobility training on functionality in children with cerebral palsy: study protocol for a double-blind randomized controlled clinical trial. BMC Pediatr. 2013 Oct 11;13:168. doi: 10.1186/1471-2431-13-168. PMID 24112817
- [Background] Volpato C, Piccione F, Cavinato M, Duzzi D, Schiff S, Foscolo L, Venneri A. Modulation of affective symptoms and resting state activity by brain stimulation in a treatment-resistant case of obsessive-compulsive disorder. Neurocase. 2013 Aug;19(4):360-70. doi: 10.1080/13554794.2012.667131. Epub 2012 May 4. PMID 22554168
- [Background] Clarkson AN, Huang BS, Macisaac SE, Mody I, Carmichael ST. Reducing excessive GABA-mediated tonic inhibition promotes functional recovery after stroke. Nature. 2010 Nov 11;468(7321):305-9. doi: 10.1038/nature09511. Epub 2010 Nov 3. PMID 21048709
- [Background] Filho PR, Vercelino R, Cioato SG, Medeiros LF, de Oliveira C, Scarabelot VL, Souza A, Rozisky JR, Quevedo Ada S, Adachi LN, Sanches PR, Fregni F, Caumo W, Torres IL. Transcranial direct current stimulation (tDCS) reverts behavioral alterations and brainstem BDNF level increase induced by neuropathic pain model: Long-lasting effect. Prog Neuropsychopharmacol Biol Psychiatry. 2016 Jan 4;64:44-51. doi: 10.1016/j.pnpbp.2015.06.016. Epub 2015 Jul 7. PMID 26160698
- [Background] Fritsch B, Reis J, Martinowich K, Schambra HM, Ji Y, Cohen LG, Lu B. Direct current stimulation promotes BDNF-dependent synaptic plasticity: potential implications for motor learning. Neuron. 2010 Apr 29;66(2):198-204. doi: 10.1016/j.neuron.2010.03.035. PMID 20434997
- [Background] Serre F, Fatseas M, Denis C, Swendsen J, Auriacombe M. Predictors of craving and substance use among patients with alcohol, tobacco, cannabis or opiate addictions: Commonalities and specificities across substances. Addict Behav. 2018 Aug;83:123-129. doi: 10.1016/j.addbeh.2018.01.041. Epub 2018 Feb 2. PMID 29428330
- [Background] Coles AS, Kozak K, George TP. A review of brain stimulation methods to treat substance use disorders. Am J Addict. 2018 Mar;27(2):71-91. doi: 10.1111/ajad.12674. Epub 2018 Feb 19. PMID 29457674
- [Background] Gladwin TE, den Uyl TE, Fregni FF, Wiers RW. Enhancement of selective attention by tDCS: interaction with interference in a Sternberg task. Neurosci Lett. 2012 Mar 14;512(1):33-7. doi: 10.1016/j.neulet.2012.01.056. Epub 2012 Feb 2. PMID 22327036
- [Background] Fregni F, Boggio PS, Nitsche M, Bermpohl F, Antal A, Feredoes E, Marcolin MA, Rigonatti SP, Silva MT, Paulus W, Pascual-Leone A. Anodal transcranial direct current stimulation of prefrontal cortex enhances working memory. Exp Brain Res. 2005 Sep;166(1):23-30. doi: 10.1007/s00221-005-2334-6. Epub 2005 Jul 6. PMID 15999258
- [Background] Dockery CA, Hueckel-Weng R, Birbaumer N, Plewnia C. Enhancement of planning ability by transcranial direct current stimulation. J Neurosci. 2009 Jun 3;29(22):7271-7. doi: 10.1523/JNEUROSCI.0065-09.2009. PMID 19494149
- [Background] Fecteau S, Pascual-Leone A, Zald DH, Liguori P, Theoret H, Boggio PS, Fregni F. Activation of prefrontal cortex by transcranial direct current stimulation reduces appetite for risk during ambiguous decision making. J Neurosci. 2007 Jun 6;27(23):6212-8. doi: 10.1523/JNEUROSCI.0314-07.2007. PMID 17553993
- [Background] Goldstein RZ, Volkow ND. Dysfunction of the prefrontal cortex in addiction: neuroimaging findings and clinical implications. Nat Rev Neurosci. 2011 Oct 20;12(11):652-69. doi: 10.1038/nrn3119. PMID 22011681
- [Background] Boggio PS, Sultani N, Fecteau S, Merabet L, Mecca T, Pascual-Leone A, Basaglia A, Fregni F. Prefrontal cortex modulation using transcranial DC stimulation reduces alcohol craving: a double-blind, sham-controlled study. Drug Alcohol Depend. 2008 Jan 1;92(1-3):55-60. doi: 10.1016/j.drugalcdep.2007.06.011. Epub 2007 Jul 19. PMID 17640830
- [Background] den Uyl TE, Gladwin TE, Wiers RW. Transcranial direct current stimulation, implicit alcohol associations and craving. Biol Psychol. 2015 Feb;105:37-42. doi: 10.1016/j.biopsycho.2014.12.004. Epub 2014 Dec 23. PMID 25541515
- [Background] Bari A, Robbins TW. Inhibition and impulsivity: behavioral and neural basis of response control. Prog Neurobiol. 2013 Sep;108:44-79. doi: 10.1016/j.pneurobio.2013.06.005. Epub 2013 Jul 13. PMID 23856628
- [Background] Dalley JW, Everitt BJ, Robbins TW. Impulsivity, compulsivity, and top-down cognitive control. Neuron. 2011 Feb 24;69(4):680-94. doi: 10.1016/j.neuron.2011.01.020. PMID 21338879
- [Background] Fineberg NA, Potenza MN, Chamberlain SR, Berlin HA, Menzies L, Bechara A, Sahakian BJ, Robbins TW, Bullmore ET, Hollander E. Probing compulsive and impulsive behaviors, from animal models to endophenotypes: a narrative review. Neuropsychopharmacology. 2010 Feb;35(3):591-604. doi: 10.1038/npp.2009.185. Epub 2009 Nov 25. PMID 19940844
- [Background] Lawrence AJ, Luty J, Bogdan NA, Sahakian BJ, Clark L. Problem gamblers share deficits in impulsive decision-making with alcohol-dependent individuals. Addiction. 2009 Jun;104(6):1006-15. doi: 10.1111/j.1360-0443.2009.02533.x. PMID 19466924
- [Background] Moreno M, Estevez AF, Zaldivar F, Montes JM, Gutierrez-Ferre VE, Esteban L, Sanchez-Santed F, Flores P. Impulsivity differences in recreational cannabis users and binge drinkers in a university population. Drug Alcohol Depend. 2012 Aug 1;124(3):355-62. doi: 10.1016/j.drugalcdep.2012.02.011. Epub 2012 Mar 15. PMID 22425410
- [Background] Gilmore CS, Dickmann PJ, Nelson BG, Lamberty GJ, Lim KO. Transcranial Direct Current Stimulation (tDCS) paired with a decision-making task reduces risk-taking in a clinically impulsive sample. Brain Stimul. 2018 Mar-Apr;11(2):302-309. doi: 10.1016/j.brs.2017.11.011. Epub 2017 Nov 22. PMID 29174303
- [Background] Shen B, Yin Y, Wang J, Zhou X, McClure SM, Li J. High-definition tDCS alters impulsivity in a baseline-dependent manner. Neuroimage. 2016 Dec;143:343-352. doi: 10.1016/j.neuroimage.2016.09.006. Epub 2016 Sep 6. PMID 27608604
- [Background] Saba G, Moukheiber A, Pelissolo A. Transcranial cortical stimulation in the treatment of obsessive-compulsive disorders: efficacy studies. Curr Psychiatry Rep. 2015 May;17(5):36. doi: 10.1007/s11920-015-0571-3. PMID 25825002
- [Background] Senco NM, Huang Y, D'Urso G, Parra LC, Bikson M, Mantovani A, Shavitt RG, Hoexter MQ, Miguel EC, Brunoni AR. Transcranial direct current stimulation in obsessive-compulsive disorder: emerging clinical evidence and considerations for optimal montage of electrodes. Expert Rev Med Devices. 2015 Jul;12(4):381-91. doi: 10.1586/17434440.2015.1037832. Epub 2015 May 17. PMID 25982412
- [Background] Val-Laillet D, Aarts E, Weber B, Ferrari M, Quaresima V, Stoeckel LE, Alonso-Alonso M, Audette M, Malbert CH, Stice E. Neuroimaging and neuromodulation approaches to study eating behavior and prevent and treat eating disorders and obesity. Neuroimage Clin. 2015 Mar 24;8:1-31. doi: 10.1016/j.nicl.2015.03.016. eCollection 2015. PMID 26110109
- [Background] Gandiga PC, Hummel FC, Cohen LG. Transcranial DC stimulation (tDCS): a tool for double-blind sham-controlled clinical studies in brain stimulation. Clin Neurophysiol. 2006 Apr;117(4):845-50. doi: 10.1016/j.clinph.2005.12.003. Epub 2006 Jan 19. PMID 16427357
- [Background] Marteau TM, Bekker H. The development of a six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI). Br J Clin Psychol. 1992 Sep;31(3):301-6. doi: 10.1111/j.2044-8260.1992.tb00997.x. PMID 1393159
- [Background] Bobes García J, G.-Portilla MP, Bascarán Fernández MT, Saiz Martínez PA, Bousoño García M. Banco de instrumentos básicos para la práctica de la psiquiatría clínica. Ars Médica, Barcelona. 2004.
- [Background] Whisman MA, Richardson ED. Normative Data on the Beck Depression Inventory--Second Edition (BDI-II) in College Students. J Clin Psychol. 2015 Sep;71(9):898-907. doi: 10.1002/jclp.22188. Epub 2015 May 7. PMID 25950150
- [Background] Stanford MS, Mathias CW, Dougherty DM, Lake SL, Anderson NE, Patton JH. Fifty years of the Barratt Impulsiveness Scale: An update and review. Personality and Individual Differences. 2009; 47(5): 385-395.
- [Background] Hodgson RJ, Rachman S. Obsessional-compulsive complaints. Behav Res Ther. 1977;15(5):389-95. doi: 10.1016/0005-7967(77)90042-0. No abstract available. PMID 612339
- [Background] Sanchez-Kuhn A, Leon JJ, Gongora K, Perez-Fernandez C, Sanchez-Santed F, Moreno M, Flores P. Go/No-Go task performance predicts differences in compulsivity but not in impulsivity personality traits. Psychiatry Res. 2017 Nov;257:270-275. doi: 10.1016/j.psychres.2017.07.064. Epub 2017 Jul 31. PMID 28783574
- [Background] Hochman S, Henik A, Kalanthroff E. Stopping at a red light: Recruitment of inhibitory control by environmental cues. PLoS One. 2018 May 3;13(5):e0196199. doi: 10.1371/journal.pone.0196199. eCollection 2018. PMID 29723204